CLINICAL TRIAL: NCT06499350
Title: A Dose-Escalation and Dose-Expansion Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of AXL Inhibitor FC084CSA Tablets in Combination With Tislelizumab in the Treatment of Advanced Malignant Solid Tumors
Brief Title: A Study of FC084CSA in Combination of Tislelizumab in Patients With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FindCure Biosciences (ZhongShan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FC084-CA-102
Record Dates: First submitted 2024-07-08; First posted 2024-07-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Intervention Model Description: FC084CSA in combination with Tislelizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FC084CSA+Tislelizumab (Experimental): This is a single arm phase I trial in a 3 + 3 dose escalation and cohort expansion design evaluating the safety and tolerability of FC084CSA in combination with Tislelizumab. Increasing dose levels of FC084CSA with fixed dose of Tislelizumab. Dose escalation continues until dose-limiting toxicities (DLT) are observed in one-third of participants. If no DLT occurs, the next cohort will be enrolled at the next planned dose level. If 1 DLT occurs in a cohort, another 3 patients will be treated with the same dose level. Following the definition of the recommended Phase 2 Dose (RP2D) of FC084CSA in dose escalation phase, NSCLC dose expansion cohort is planned to perform a preliminary assessment of the anti-tumour efficacy and to further establish the safety profile of the RP2D of FC084CSA in combination with Tislelizumab.
  Interventions: Drug: FC084CSA+Tislelizumab combination (dose escalation); Drug: RP2D of FC084CSA+Tislelizumab combination (dose expansion)

INTERVENTIONS:
Drug: FC084CSA+Tislelizumab combination (dose escalation) — Increasing dose levels of FC084CSA+fixed dose Tislelizumab combination therapy
  Other Names: FC084CSA+BGB-A317 combination (dose escalation)
Drug: RP2D of FC084CSA+Tislelizumab combination (dose expansion) — RP2D of FC084CSA+fixed dose Tislelizumab combination therapy
  Other Names: RP2D of FC084CSA+BGB-A317 combination (dose expansion)

SUMMARY:
The goal of this clinical trial is to learn the safety, tolerability, pharmacokinetic characteristics and efficacy of FC084CSA in combination with Tislelizumab in patients with advanced malignant solid tumors.

DETAILED DESCRIPTION:
The study includes two phases. Phase Ib adopts a "3+3" dose escalation design to assess safety and tolerability of increasing dose levels of FC084CSA in combination of fixed dose of Tislelizumab. Phase IIa is the dose expansion phase to further observe the preliminary effectiveness of the recommended Phase 2 Dose of FC084CSA in combination of Tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old male and female.
2. Phase Ib: Patients with histologically or cytologically diagnosed solid tumors who have failed standard therapy; Phase IIa: Patients with histologically or cytologically confirmed stage IIIB/IIIC and stage IV NSCLC which surgery or radiotherapy cannot be performed.
3. No known sensitizing mutations or other actionable oncogenes with approved therapies if available.
4. Prior PD-1/PD-L1 inhibitor combined with platinum-containing therapy failed;
5. According to RECIST 1.1, there is at least one measurable lesion.
6. ECOG performance status 0-1.
7. Major organs are functioning well.

Exclusion Criteria:

1. Not recovered from the adverse reactions caused by previous anti-tumor treatments (≥CTCAE grade 1).
2. Received anti-tumor therapy within 4 weeks before enrollment.
3. Participated in other clinical trials within 4 weeks before enrollment and used clinical investigational drugs during this period.
4. Have undergone surgery within 4 weeks before enrollment, and the investigator believes that the patient's state has not recovered to the point where the study can be started.
5. Patients with ascites (ascites), pleural effusion (pleural effusion) or pericardial effusion that cannot be controlled by drainage or other methods.
6. Central nervous system metastases with clinical symptoms.
7. With any situations that the researcher considers inappropriate to participate in this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) | Approximately 8 months
  The highest dose is defined at which no more than 1 of 3 evaluable participants has had a Dose Limiting Toxicity (DLT) according to NCI CTCAE V5.0 criteria and determination by Investigator and Data and Safety Monitoring Committee.
Determine the Recommended Phase 2 Dose (RP2D) | Approximately 8 months
  The RP2D is based upon the review of all available data including safety, pharmacokinetic, preliminary anti-tumor activity, and MTD.
Determine dose-limiting toxicity (DLT) | 21 days after first dose
  Determine the DLT of FC084CSA
Objective response rate (ORR) | Approximately 12 months
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Approximately 12 months
  DCR as assessed using RECIST 1.1
Progression free survival (PFS) | Approximately 12 months
  PFS as assessed using RECIST 1.1
Overal suvival (OS) | Approximately 18 months
  It is defined as the time from date of first dose to the date of death (due to any cause). Subjects who are alive will be censored at the last known alive dates.
Pharmacokinetic (PK) Cmax | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) Tmax | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) AUC 0-t | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) AUC 0-∞ | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No